CLINICAL TRIAL: NCT06628999
Title: Perceptual-vision Training As a Strategy for Healthy Ageing in Adults with Intellectual Disability
Brief Title: Perceptual-vision Training and Intellectual Disabilities
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Luca Cavaggioni, Principal Investigator, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0119168
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-10

CONDITIONS: Intellectual Disability; Intellectual Impairment; Activity, Motor; Sports Physical Therapy
Keywords: Visual training; Intellectual disability; Physical activity
MeSH Terms: conditions — Intellectual Disability; Motor Activity | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Visual Training Group (Experimental): Visual Training Group: physical training exercises aiming to combine visual skills with basic motor actions for 16 consecutive weeks
  Interventions: Other: Visual Training
- Control Group (Active Comparator): Control Group: active lifestyle based on healthy habits for 16 consecutive weeks
  Interventions: Other: Control Group
- Visual Training-detraining Group (Experimental): Visual Training-detraining Group: physical exercises physical training exercises aiming to combine visual skills with basic motor actions for 8 consecutive weeks. The last remaining 8 weeks (up to 16 week) the group will conduct a period of detraining in which no physical exercises will be administered
  Interventions: Other: Visual Training-detraining

INTERVENTIONS:
Other: Visual Training — 16-week training protocol focused on visual training designed for ameliorating cognitive performance and physical fitness
  Arms: Visual Training Group
Other: Control Group — 16-week of active lifestyle based on healthy habits
  Arms: Control Group
Other: Visual Training-detraining — 8-week training protocol focused on visual training designed for ameliorating cognitive performance and physical fitness, followed by 8 week with no specific training protocol
  Arms: Visual Training-detraining Group

SUMMARY:
Physical activity for healthy ageing is an important feature and the possibility to detect practical solutions to solve the need for feasible health promotion interventions to reduce health disparities and wellbeing in individuals with intellectual disability (ID) is an open question. In this perspective, vision has a remarkable role in spatial cognition and organization, especially in individuals with ID. Therefore, the aim is to investigate the effectiveness of a perceptual-vision training program on cognitive performance (inhibitory control) and physical fitness (balance, agility and muscular strength) in adults with ID throughout 16 weeks. Participants with mild ID will be randomly divided into a perceptual-vision training group, a perceptual-vision training-detraining group and a control group. Cognitive performance and physical fitness will be assessed at baseline, mid and at the end of 16 weeks. In conclusion, a visual training program may present the potentiality to impact various health domains, from cognition to physical performance in individuals with intellectual disabilities, promoting their healthy aging.

DETAILED DESCRIPTION:
Despite the importance of physical activity for healthy ageing and the need for feasible health promotion interventions to reduce health disparities and improve aging wellbeing in individuals with intellectual disability (ID), there is a lack of empirically supported strategies for health promotion and disease prevention in adults with ID. Notably, vision and eye tracking play a key role in spatial cognition and orientation triggering several brain areas and people with ID may present anomalous visual movements, spatial organization or cognitive performance. The aim of the present project is to investigate a potential strategy for promoting healthy ageing targeting both physical and cognitive domains in individuals with ID. Specifically, this project will study the effect of a perceptual-vision training program on cognitive performance (inhibitory control) and physical fitness (balance, agility and muscular strength) in adults with ID. The second aim is to test the association between cognitive and physical performance variables. Participants with mild ID will be randomly allocated to a perceptual-vision training group (n = 28), a perceptual-vision training-detraining group (n = 28) and a control group (n = 28).

During the overall 16 weeks, the perceptual-vision training group will follow an intervention protocol based on vision and oculomotor exercises combined with balance motor actions for the entire period, the perceptual-vision training-detraining group will follow the same oculomotor training program for 8 weeks and a period of detraining for the last consecutive 8 weeks. Lastly, the control group will continue to perform habitual active lifestyle for 16 weeks. Cognitive performance and physical fitness will be assessed at baseline, mid (end of 8 week), and post intervention period (end of 16 week). Overall, a perceptual-vision training program may have the potential to positively impact various aspects of life quality in individuals with ID promoting autonomy, health, social integration, and overall wellbeing. This may be a promising strategy to ameliorate healthy ageing of people with ID across various domains.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 70 years
* mild ID (Intellectual Quotient = 51-69).

Exclusion Criteria:

* inability to understand basic verbal communication
* strict dependence on personnel or assistive support devices
* presence of concomitant sensorial or physical impairments
* presence of behavioural problems or any other clinical condition that may compromise the regular physical activity practice

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2025-10-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline cognitive performance at 16 week | Up to sixteen weeks
  Response time on a computerized test conceptualized as a measure of cognitive performance inhibitory control (Modified Flanker Task test). Participants are tasked with identifying the direction of the central target stimulus that is flanked by either congruent (<<<<<) or incongruent (>><>>) stimuli by pressing the correct keyboard key.

SECONDARY OUTCOMES:
Change from baseline static balance at 16 week | Up to sixteen weeks
  Postural control detected in standing position with eyes closed using the Balance Error Scoring System protocol in arbitrary units using a 0-30 point scale in which lower scores mean a better outcome result
Change from baseline strength at 16 week | Up to sixteen weeks
  Maximal isometric grip in kilograms using the handgrip dynamometer
Change from baseline strength at 16 week | Up to sixteen weeks
  Amount of time in seconds during a chair rise for five consecutive times adopting the Five Repetition sit to stand test
Change from baseline movement agility at 16 week | Up to sixteen weeks
  Amount of time in seconds using the Time Up and Go test. The test begins with the participant that should stand up from a chair, he has to walk forward for three meters, then to come back and to sit down on a chair. During the entire procedure the participant should count backward by three starting from a casual number

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cavaggioni, PhD, Principal Investigator — Universitià degli Studi dell'Insubria

REFERENCES:
- [Background] Carmeli E, Imam B. Health promotion and disease prevention strategies in older adults with intellectual and developmental disabilities. Front Public Health. 2014 Apr 14;2:31. doi: 10.3389/fpubh.2014.00031. eCollection 2014. PMID 24783190
- [Background] Erickson KI, Hillman C, Stillman CM, Ballard RM, Bloodgood B, Conroy DE, Macko R, Marquez DX, Petruzzello SJ, Powell KE; FOR 2018 PHYSICAL ACTIVITY GUIDELINES ADVISORY COMMITTEE*. Physical Activity, Cognition, and Brain Outcomes: A Review of the 2018 Physical Activity Guidelines. Med Sci Sports Exerc. 2019 Jun;51(6):1242-1251. doi: 10.1249/MSS.0000000000001936. PMID 31095081
- [Background] Formenti D, Duca M, Trecroci A, Ansaldi L, Bonfanti L, Alberti G, Iodice P. Perceptual vision training in non-sport-specific context: effect on performance skills and cognition in young females. Sci Rep. 2019 Dec 10;9(1):18671. doi: 10.1038/s41598-019-55252-1. PMID 31822740
- [Background] Forte R, Trentin C, Tocci N, Lucia S, Aydin M, Di Russo F. Motor-cognitive exercise with variability of practice and feedback improves functional ability and cognition in older individuals. Aging Clin Exp Res. 2023 Nov;35(11):2797-2806. doi: 10.1007/s40520-023-02568-8. Epub 2023 Oct 19. PMID 37853304
- [Background] Giuliani F, Favrod J, Grasset F, Schenk F. Accurate memory for object location by individuals with intellectual disability: absolute spatial tagging instead of configural processing? Res Dev Disabil. 2011 May-Jun;32(3):986-94. doi: 10.1016/j.ridd.2011.01.055. Epub 2011 Feb 24. PMID 21353464
- [Background] Henderson JM. Human gaze control during real-world scene perception. Trends Cogn Sci. 2003 Nov;7(11):498-504. doi: 10.1016/j.tics.2003.09.006. PMID 14585447
- [Background] Horner-Johnson W, Bailey D. Assessing Understanding and Obtaining Consent from Adults with Intellectual Disabilities for a Health Promotion Study. J Policy Pract Intellect Disabil. 2013 Sep;10(3):10.1111/jppi.12048. doi: 10.1111/jppi.12048. PMID 24223054
- [Background] Krahn GL, Fox MH. Health disparities of adults with intellectual disabilities: what do we know? What do we do? J Appl Res Intellect Disabil. 2014 Sep;27(5):431-46. doi: 10.1111/jar.12067. Epub 2013 Jul 31. PMID 23913632
- [Background] Santos FH, Zurek J, Janicki MP. Efficacy of Healthy Aging Interventions for Adults With Intellectual and Developmental Disabilities: A Systematic Review. Gerontologist. 2022 Apr 20;62(4):e235-e252. doi: 10.1093/geront/gnaa192. PMID 33220058
- [Background] Wollesen B, Wildbredt A, van Schooten KS, Lim ML, Delbaere K. The effects of cognitive-motor training interventions on executive functions in older people: a systematic review and meta-analysis. Eur Rev Aging Phys Act. 2020 Jul 2;17:9. doi: 10.1186/s11556-020-00240-y. eCollection 2020. PMID 32636957
- [Derived] Cavaggioni L, Formenti D, Castiglioni P, Ardigo LP, Merati G. Perceptual-vision training as a strategy for healthy aging in adults with intellectual disability: a study protocol. Front Psychol. 2025 Apr 24;16:1526826. doi: 10.3389/fpsyg.2025.1526826. eCollection 2025. PMID 40342338